CLINICAL TRIAL: NCT00661336
Title: An Open-Label, Multicenter, Phase 1 Dose Escalation Study to Evaluate Safety, Tolerability and Anti-tumor Activity of Systemic Buthionine Sulfoximine (BSO) in Combination With Normothermic Isolated Limb Infusion of Melphalan in Subjects With Locally Advanced In-Transit Malignant Melanoma
Brief Title: A Phase I Trial of Normothermic Isolated Limb Infusion (ILI) With Melphalan Plus Buthionine Sulfoximine (BSO) in Patients With Locally Advanced Malignant Melanoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was withdrawn due to lack of patients.
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: Pro00001793; DUMC-PRO00001793 (Other: NCI CDR0000592735)
Record Dates: First submitted 2008-04-17; First posted 2008-04-18 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2010-04

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Buthionine Sulfoximine; Melphalan; Microarray Analysis; Chromatography, High Pressure Liquid; Biopsy

INTERVENTIONS:
Drug: buthionine sulfoximine
Drug: melphalan
Genetic: microarray analysis
Other: high performance liquid chromatography
Other: laboratory biomarker analysis
Other: pharmacological study
Procedure: biopsy

SUMMARY:
RATIONALE: Buthionine sulfoximine may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as melphalan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Sometimes when chemotherapy is given, it does not stop the growth of tumor cells. The tumor is said to be resistant to chemotherapy. Giving buthionine sulfoximine together with chemotherapy may reduce drug resistance and allow the tumor cells to be killed.

PURPOSE: This phase I trial is studying the side effects and best dose of melphalan when given as an isolated limb infusion together with buthionine sulfoximine in treating patients with persistent or recurrent stage III malignant melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose of melphalan when administered as an isolated limb infusion in combination with a systemic infusion of buthionine sulfoximine (BSO) in patients with persistent or recurrent stage IIIB or IIIC in-transit malignant melanoma.

Secondary

* To define the dose-limiting toxicity of regional melphalan when administered with systemic BSO in these patients.
* To determine whether the combination of systemic BSO and regional melphalan can yield clinical responses in patients who have not responded well to prior melphalan-based regional treatment.
* To determine the effectiveness of systemic BSO in decreasing tumor glutathione (GSH) levels and its effect on GST activity and GST expression.
* To examine the correlation between tumor GSH levels and GSH levels in peripheral blood mononuclear cells to determine if the latter can serve as a surrogate marker for tumor GSH depletion.
* To determine the pharmacokinetics of systemic BSO and regional melphalan in these patients.
* To determine if BSO alters the mRNA expression signature of melphalan resistance.
* To determine, preliminarily, the efficacy of systemic BSO and regional melphalan in these patients.
* To correlate baseline mRNA expression signature of melphalan resistance with treatment efficacy.

OUTLINE: This is a multicenter, dose-escalation study of melphalan.

Patients receive buthionine sulfoximine (BSO) IV continuously on days 1-3 and melphalan as an isolated limb infusion (ILI) over 30 minutes on day 2 in the absence of progressive disease or unacceptable toxicity.

Patients undergo biopsies and blood sample collection at baseline, immediately before and during ILI, and then at 12 weeks after ILI or at the time of disease progression. Samples are analyzed for GST genotype, tumor glutathione (GSH) levels (by enzymatic assay or HPLC/fluorescence detection [FLD]), drug pharmacokinetics, and mRNA expression signature of melphalan resistance.

After completion of study treatment, patients are followed at 2, 6, and 12 weeks, every 3 months for 1 year, and then every 6 months for up to 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven primary or recurrent in-transit melanoma of the extremity

  * Stage IIIB or IIIC disease, as determined by whole body imaging with a CT scan of the chest, abdomen, and pelvis AND PET scan within the past 4 weeks

    * Patients with stage IIIC disease must have undergone removal of regional lymph nodes
    * Patients with indeterminate staging must be reviewed by the study chairs prior to study registration
* Previously treated with melphalan-based regional therapy and had persistent disease at 3 months OR achieved a complete response but disease recurred within 6 months
* Disease to be treated by regional therapy must be distal to the planned site of tourniquet placement
* Bidimensionally measurable disease by caliper or a radiological method as defined by the RECIST criteria modified for cutaneous lesions

  * Photo documentation required
  * Patients with a single lesion must have archived tumor tissue available for study analysis
* No history of tumors with clinically significant evidence of active bleeding (e.g., gross hemoptysis, hematemesis, hematuria, melena, or bleeding superficial tumor) within the past 12 weeks
* No stage IV disease
* No cerebral metastases

PATIENT CHARACTERISTICS:

* ECOG/Zubrod performance status 0-1
* Serum creatinine ≤ 1.5 mg/dL
* WBC ≥ 3,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL
* Bilirubin normal
* AST and ALT ≤ 2.5 times normal
* Must have a palpable femoral/axillary pulse in the affected extremity
* No uncontrolled seizures or clinically significant CNS disorders
* No psychiatric condition or diminished capacity that could preclude study compliance or giving informed consent
* No history of allergic reactions and/or hypersensitivity to melphalan
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of other malignancies except adequately treated basal cell or squamous cell carcinoma of the skin; curatively treated carcinoma in situ of the uterine cervix, prostate cancer, or superficial bladder cancer; or other curatively treated solid tumors with no evidence of disease for ≥ 5 years
* No stroke or other major tissue injury within the past 4 weeks
* No other uncontrolled serious chronic disease or condition that, in the investigator's opinion, could preclude study compliance or follow-up

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* More than 4 weeks since prior major surgery

  * Wound healing adequate since last major surgery
* More than 4 weeks since prior antineoplastic therapy, radiotherapy, or any other investigational drug
* More than 7 days since prior antimicrobial agents (i.e., antibiotic, antifungal, or antiviral agents) for active infection or infectious symptoms
* No drugs that are known to cause enhanced glutathione depletion (e.g., acetaminophen) for 7 days before, during, and for 7 days after buthionine sulfoximine (BSO) administration
* No cephalosporin antibiotics for 7 days before, during, and for 7 days after BSO administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of melphalan when administered as an isolated limb infusion in combination with a systemic infusion of buthionine sulfoximine (BSO)

SECONDARY OUTCOMES:
Dose-limiting toxicity of regional melphalan when administered with systemic BSO
Clinical response
Effectiveness of systemic BSO in decreasing tumor glutathione (GSH) levels and its effect on GST activity and GST expression
Correlation between tumor GSH levels and GSH levels in peripheral blood mononuclear cells to determine if the latter can serve as a surrogate marker for tumor GSH depletion
Pharmacokinetics
mRNA expression signature of melphalan resistance
Efficacy as defined by the RECIST criteria modified for cutaneous lesions
Correlation of baseline mRNA expression signature of melphalan resistance with treatment efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Douglas S. Tyler, MD, Principal Investigator — Duke Cancer Institute
Locations (2):
- United States (2):
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas